CLINICAL TRIAL: NCT03539289
Title: An Open Label Phase IV, Multicenter, International, Interventional Study to Evaluate the Effect of Diet on Gastrointestinal Adverse Events in Patients With IPF Treated With Pirfenidone
Brief Title: Evaluate the Effect of Diet on Gastrointestinal Adverse Events in Patients With IPF Treated With Pirfenidone
Acronym: MADIET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government)
Collaborators: Institut d'Investigació Biomèdica de Bellvitge (Other); Hospital Universitari de Bellvitge (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA39293-DIET; 2016-003827-45 (EudraCT Number)
Record Dates: First submitted 2018-05-16; First posted 2018-05-29 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Pulmonary Disease
Keywords: IPF; Mitigating Adverse Events
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MUFA Diet (Other): Monounsaturated Fatty Acids Diet
  Interventions: Behavioral: MUFA Diet
- SFA Diet (Other): Saturated Fatty Acids Diet
  Interventions: Behavioral: SFA Diet

INTERVENTIONS:
Behavioral: MUFA Diet — Control of patient MUFA Diet
  Arms: MUFA Diet
Behavioral: SFA Diet — Control of patient SFA Diet
  Arms: SFA Diet

SUMMARY:
The primary objective is to compare the incidence of gastrointestinal AEs in patients treated with IPF, initiating pirfenidone for the first time, according to the type of diet (MUFA vs SFA). Gastrointestinal AEs rates between study groups will be evaluated during the first 16 weeks of pirfenidone treatment.

DETAILED DESCRIPTION:
IPF is a chronic, progressive, irreversible disease that ends in respiratory failure and death. The average survival time is 2-5 years from the onset of the first symptoms. IPF patients are often treated with pirfenidone, and the response is positive, however there are gastrointestinal side effects. The data published about patient adherence to pirfenidone treatment relates to the emergence of gastrointestinal AEs, which is variable and appears to have a lower incidence in the hospitals in the south of Europe, who report fewer serious gastrointestinal AEs than in countries from the north of Europe.

Recent data from the Spanish Registry have reported a prevalence of 6,3% of GI effects with pirfenidone in 270 IPF patients under treatment (IPF-Spanish Registry June 2016), while in Netherlands and Belgium the reported GI effects are around 36%, and associated with treatment discontinuation in 7,9% of patients.

Even though the ingestion of food during the taking of medication and other measures recommended for the prevention of symptoms may have a beneficial effect with respect to gastrointestinal AEs, up to now there have been no studies about the influence of diet on these events. Therefore, it is possible that the differences in the patients' habitual diet, i.e. the composition in quantity and types of fat ingested, may be the source of the variability of the gastrointestinal AEs observed between countries.

Distinct dietary models have been taking shape over the past decades. In countries such as England, central and northern Europe, and a large part of North America, dietary habits characterized by a high consumption of saturated and hydrogenated fats in the form of pastries and pre-cooked products, veal, pork, and lamb (>150 g per day), butter and milk fats, and scant consumption of fruits, greens, vegetables, and whole-grain cereals. It is called the Occidental Diet (OD). Various studies have associated it, as an environmental factor, with diseases such as vascular accidents, diabetes, metabolic syndrome, and various types of cancer.

On the other hand, traditional Mediterranean diets have been associated with low rates of chronic diseases and high life expectancy among the populations that consume them. They are characterized by an abundance of greens, garden produce, fresh fruit, legumes and cereals; a variable quantity, according to the zone, of olive oil, which is the main cooking fat; a moderate consumption of alcohol, mainly in the form of wine; some fish; moderate ingestion of dairy foods, and low consumption of meat.

The main characteristic of the Mediterranean diet is that the ratio of monounsaturated fatty acids (MUFA) to saturated fatty acids (SFA) is much higher than in other zones of Europe and North America due to a high consumption of olive oil as the main cooking oil. Olive oil fills distinct functions in the gastrointestinal tract. Being the fat that provides the best digestibility and whose mechanism of action is based on an inhibition of gastric motility, thus promoting a lower degree of gastroesophageal reflux. That is the reason that it is used extensively among Nutrition professionals when patients present low oral tolerance(22-24). Olive oil, also, has been used to mitigate postoperative nausea and vomiting.

This study will analyze the AEs in IPF patients in 6 countries, who are prescribed pirfenidone. They will be divided into SFA and MUFA arms and the AEs of each arm statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Ability to comply with the study protocol in the opinion of the Investigator
* Age > 40 years
* Naiive-treated patients with diagnosis of IPF at least 1 week but not more than 5 years prior to study baseline
* Confirmation of IPF diagnosis by the Investigator of each Centre, in accordance with the 2011 international consensus guidelines (Raghu et al. 2011), at baseline
* IPF that meet criteria for pirfenidone treatment initiation according to local reimbursement policy
* Approval of potential study participation by Central Committee (FFQ shows a clear diet predominance).

Defined and regular diet for at least six months prior to baseline (i.e. no frequent changes in the type of diet).

* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use a non-hormonal contraceptive method with a failure rate of <1% per year during the Treatment Period and for at least 28 days after the last dose of study treatment
* For men who are not surgically sterile: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm

Exclusion Criteria:

* • History of coexistent and clinically significant (in the opinion of the Investigator) chronic obstructive pulmonary disease (COPD), bronchiectasis, asthma, inadequately treated sleep-disordered breathing, or any clinically significant pulmonary diseases or disorders other than IPF

  * History of any connective tissue disease, including, but not limited to: rheumatoid arthritis, scleroderma, polymyositis/dermatomyositis, systemic lupus erythematosus, or mixed connective tissue disease
  * History of clinically significant environmental exposure to agents known to cause pulmonary fibrosis, including asbestos, beryllium, silica, and other occupational dusts; amiodarone, nitrofurantoin, and other drugs; radiation; and birds, feathers, molds, and other inhaled antigens known to cause hypersensitivity pneumonitis
  * Participation in any other investigational trial throughout the study
  * Any serious medical condition that, in the opinion of the Investigator, may pose an additional risk in administering study treatment to the patient
  * Expecting a lung transplant in <12 months
  * Certain laboratory abnormalities or findings at baseline, including:

    * Total bilirubin > 5 the upper limit of normal (ULN)
    * AST/SGOT or ALT/SGPT >1.5 ULN
    * Alkaline phosphatase >2.0 ULN
    * Creatinine clearance <40 mL/min, calculated using the Cockcroft-Gault formula
  * Pregnant or lactating, or intending to become pregnant during the study
  * Pharmacological treatments (concomitant-therapy) at baseline that may cause patient gastrointestinal side effects
  * Major gastro-intestinal disorders at baseline (gastric or bowel surgery, ulcus). Patients with gastroesophagic reflux or other minor digestive disorders can be included.
  * Pregnant patients, or women of child-bearing potential, not using a reliable non-hormonal? contraceptive method
  * Planning to change the type of diet in the next 4 months
  * Not able to follow a specific type of diet or cannot be allocated to a specific type of diet (MUFA vs SFA) by the Central Committee
  * Previous use, intolerance, or allergy to pirfenidone or hypersensitivity to the active substance or to any of the excipients

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-12-28 (Actual); Primary Completion 2020-04-22 (Actual); Study Completion 2020-04-22 (Actual)

PRIMARY OUTCOMES:
Incidence of gastrointestinal AEs | First 16 weeks of pirfenidone treatment
  • To compare the incidence of gastrointestinal AEs in patients with IPF initiating pirfenidone for the first time - according to the type of diet (Monounsaturated Fatty Acids [MUFA] vs Saturated Fatty Acids [SFA]). Gastrointestinal AEs rates between study groups will be evaluated during the first 16 weeks of pirfenidone treatment

CONTACTS AND LOCATIONS:
Overall Officials: María Molina Molina, Principal Investigator — Unidad Funcional de Intersticio Pulmonar (UFIP).Servicio de Neumología. Hospital Universitario de Bellvitge
Locations (6):
- University Hospital Essen, Essen, Germany
- University of Crete, Eraklion, Heraklion, Greece
- Università de Catania, Catania, Sicily, Italy
- Erasmus MC, Rotterdam, Rotterdam, Netherlands
- Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain
- Brompton Hospital, London, United Kingdom

REFERENCES:
- [Derived] Molina-Molina M, Shull JG, Vicens-Zygmunt V, Rivera-Ortega P, Antoniou K, Bonella F, Renzoni E, Russell AM, Maher TM, Vancheri A, Bachs A, Aviles V, Palma J, Bermudo G, Suarez-Cuartin G, Tebe C, Rigo-Bonnin R, Montes-Worboys A, Wijsenbeek M, Vancheri C. Gastrointestinal pirfenidone adverse events in idiopathic pulmonary fibrosis depending on diet: the MADIET clinical trial. Eur Respir J. 2023 Oct 19;62(4):2300262. doi: 10.1183/13993003.00262-2023. Print 2023 Oct. PMID 37857429